CLINICAL TRIAL: NCT05962372
Title: Culturally Adapted Dietary Clinical Trial in PR: Puerto Rico Evaluation of a Culturally Informed Sustainable Intervention for Optimal Nutrition (PRECISION)
Brief Title: Culturally Adapted Dietary Clinical Trial in PR
Acronym: PRECISION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: FDI Clinical Research (Other); Yale University (Other); Broad Institute of MIT and Harvard (Other)
Responsible Party: Principal Investigator, Josiemer Mattei, Donald and Sue Pritzker Associate Professor of Nutrition, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB23-0951
Record Dates: First submitted 2023-07-14; First posted 2023-07-27 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2; Obesity; Hypertension; Dyslipidemias; High Triglycerides; High Blood Glucose; Abdominal Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Hypertension; Dyslipidemias; Hypertriglyceridemia; Hyperglycemia; Obesity, Abdominal | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be unaware of which educational messages are considered intervention or control. Investigators will not be in contact with participants and will only receive coded data. Outcome assessor will be unaware of treatment allocation of participant. Senior investigators, Research Assistants, and laboratory personnel will be blinded to the participants' group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Intervention group will receive culturally-tailored portion-control Mediterranean-like advice through monthly individual counseling for 6 months, reinforced with daily text messages for 12 months, and a monthly household supply of legumes (i.e., beans and peanuts), vegetable oils (i.e., olive oil + a blend of canola and soybean), and locally sourced assorted fruit and vegetables for 18 months. From months 18 to 24, we will monitor maintenance of behavior (no food or counseling) with support from the nutritionist available.
  Interventions: Behavioral: Culturally tailored food and diet advice
- Control (Active Comparator): Control group will receive portion-control standard non-tailored nutritional counseling in monthly individual sessions for 6 months, reinforced with daily text messages for 12 months, and monthly assistance to purchase healthy foods for 18 months. From months 18 to 24, we will monitor maintenance of behavior (no voucher or counseling), with support from the nutritionist available.
  Interventions: Behavioral: Standard healthy eating advice

INTERVENTIONS:
Behavioral: Culturally tailored food and diet advice — Puerto Rico-tailored education includes strategies for healthy eating, preferences for traditional healthy foods, recommendations for limiting unhealthy traditional foods, portion sizes, etc.
  Arms: Intervention
Behavioral: Standard healthy eating advice — Standard healthy eating education includes strategies, foods, portions, and cooking and eating tips included in the My Plate For A Healthy Puerto Rico dietary recommendations.
  Arms: Control

SUMMARY:
This project will determine whether a diet culturally adapted to adults in Puerto Rico can effectively decrease cardiometabolic risk factors. This will help define a culturally-appropriate, feasible, and sustainable diet intervention aimed at reducing cardiovascular, type 2 diabetes, and obesity outcomes.

DETAILED DESCRIPTION:
This intervention will culturally tailor a diet to the adult population in Puerto Rico based on staple foods as well as culturally appropriate strategies to reduce cardiometabolic risk factors. Based on preliminary results from studies on the island, investigators will conduct a 24-month, 2-arm intervention among 250-350 adults (125-175 per arm) ages 30-65 living in Puerto Rico with at least 1 of 5 cardiometabolic risk factors. The two arms are (1) intervention group with culturally-tailored portion-control Mediterranean Diet-like advice through monthly individual counseling for 12 months, reinforced with daily text messages for 12 months, and a monthly household supply of legumes, vegetable oils, and locally sourced assorted fruit and vegetables for 18 months; (2) control arm with portion-control standard non-tailored nutritional counseling in monthly individual sessions for 12 months, reinforced with daily text messages for 12 months, and monthly assistance to purchase healthy foods for 18 months. From months 18-24, we will monitor behavior maintenance (no food/voucher or counseling), with support from the nutritionist, and cues-to-action texts. Investigators will measure changes in cardiometabolic risk factors and metrics of eating behaviors and psychological factors. The two co-primary outcomes are changes in ASCVD score and cardiometabolic improvement score.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-65y old at the time of enrollment
2. Non-institutionalized
3. Living in PR at the time of recruitment and for at least the previous year and not planning to move from the island within the next 3 years
4. Able to answer questions without assistance
5. Having a cellphone with the capacity to receive text messages and be willing to receive daily text messages from the study on the designated cellphone number
6. Having at least one of the following:

   1. elevated BMI
   2. elevated waist circumference
   3. self-reported physician-diagnosed hypertension or use of hypertension medication or measured high blood pressure at the baseline visit
   4. self-reported physician-diagnosed pre-diabetes or measured pre-diabetes at the baseline visit
   5. self-reported physician-diagnosed dyslipidemia or use of lipid-lowering agents or laboratory values confirming dyslipidemia

Exclusion Criteria:

1. Under 30 or over 65 years of age (on the day of the interview).
2. Currently not living in Puerto Rico or not lived on the island for at least 1 year or planning to move within 3 years
3. Institutionalized
4. Not able to answer questions without assistance
5. Not having at least 1 of the five listed metabolic criteria
6. Self-reported physician-diagnosed type 1 or type 2 diabetes or use of diabetes medication (including insulin) or diabetes-diagnosis values confirmed by laboratory
7. Self-reported pregnancy
8. Gastrointestinal or chronic condition that would impact eating behaviors or nutritional status
9. Intolerance or allergies to legumes (i.e.: beans and nuts), vegetable oils (i.e.: corn, olive, canola), or fresh produce
10. Living with another person participating in the study
11. Participating in another research study that conflicts with PRECISION

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2029-05-02 (Estimated); Study Completion 2029-05-02 (Estimated)

PRIMARY OUTCOMES:
10-year risk score for a first atherosclerotic CVD event (ASCVD score) | 6; 12; 18; 24 months
  Estimate the change in first atherosclerotic CVD event (ASCVD) score; the score is calculated using the Pooled Cohort Equation which accounts for biological sex, age, race, total cholesterol, HDL-C, systolic blood pressure, treatment for high blood pressure, current diabetes diagnosis, and smoking status. Scores are expressed as percentage (0-100) with higher scores indicative of higher 10-year risk for ASCVD event. It is categorized as low-risk <5%; borderline risk 5% to 7.4%; intermediate risk 7.5% to 19.9%; and high risk ≥20%.
Cardiometabolic Improvement Score (CIS) | 6; 12; 18; 24 months
  Estimate the change in the score; calculated as the added number of risk factors changed over a predefined value; range of 0 to 10; from less to more improvement.

SECONDARY OUTCOMES:
Changes in diet quality score | 6; 12; 18; 24 months
  Determine the change in score of short diet quality screener (range 18-54; from lowest to highest quality)
Changes in diet satisfaction: diet satisfaction scale | 6; 12; 18; 24 months
  Determine the change in the score of the Diet Satisfaction Questionnaire (DSat-45) (range 45-225; from lowest to highest satisfaction) and its summed seven subscales (ranges 5-40)
Changes in intake of pre-specified food groups (fruit; vegetables; legumes; oils; meat; fat) | 6; 12; 18; 24 months
  Determine the change in servings/week of food groups
Change in levels of waist circumference | 6; 12; 18; 24 months
  Estimate the change in the value of waist circumference (cm)
Change in levels of BMI | 6; 12; 18; 24 months
  Estimate the change in the value of body mass index (kg/m2)
Change in levels of blood pressure risk factors | 6; 12; 18; 24 months
  Estimate the change in the value of systolic and diastolic blood pressure (mmHg)
Change in levels of metabolic risk factors | 6; 12; 18; 24 months
  Estimate the change in the value of glucose, triglycerides, total cholesterol, LDL, HDL (mg/dL)
Change in food security status | 6; 12; 18; 24 months
  Estimate the change in food security status assessed by the USDA Food Security Module
Change in self-efficacy score | 6; 12; 18; 24 months
  Estimate the change in self-efficacy score assessed by the Nutritional Self-Efficacy Scale

OTHER OUTCOMES:
Change in social connectedness score | 6; 12; 18; 24 months
  Estimate the change in social connectedness score from the Social Connectedness Scale/Social Assurance Scale
Change in social support score | 6; 12; 18; 24 months
  Estimate the change in social support score from the 12-item Social Support Scale

CONTACTS AND LOCATIONS:
Overall Officials: Josiemer Mattei, PhD, MPH, Principal Investigator — Harvard Chan School of Public Health; Jose F Rodriguez Orengo, PhD, Study Director — FDI Clinical Research
Locations (1):
- FDI Clinical Research, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
IPD will be managed and distributed observing NIH and IRB policies on the dissemination and sharing of research results. Study information and requests for data will be available immediately upon the data being de-identified and properly revised for quality control by contacting study investigators.
Supporting Information: Study Protocol, ICF
Time Frame: 10 years
Access Criteria: The requested data will be shared with investigators via a secured, password-protected software website, upon request.